CLINICAL TRIAL: NCT05069714
Title: Effect of One-week vs Two-week Discontinuation of Methotrexate on Efficacy of Seasonal Influenza Vaccination in Patients With Rheumatoid Arthritis: A Randomized Clinical Trial
Brief Title: One or Two Week Methotrexate Discontinuation on Efficacy of Influenza Vaccination in Rheumatoid Arthritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2109-020-1252
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis; Autoimmune Diseases; Influenza; Vaccine Reaction
Keywords: rheumatoid arthritis; methotrexate; influenza
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases; Influenza, Human

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Single-blinded study. Investigators assessing disease activity will be blinded to the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTX 1 week hold (Experimental): Patients who will hold MTX for 1 week after an influenza vaccine.
  Interventions: Drug: MTX-hold
- MTX 2 week hold (Active Comparator): Patients who will hold MTX for 2 weeks after an influenza vaccine.
  Interventions: Drug: MTX-hold

INTERVENTIONS:
Drug: MTX-hold — Temporary discontinuation of methotrexate for 1 or 2 weeks

SUMMARY:
This is a multi-center, randomized, single-blinded, prospective, parallel group intervention study to investigate whether methotrexate (MTX) discontinuation for 1 week is non-inferior to MTX discontinuation for 2 weeks in regard to satisfactory vaccination response to a seasonal influenza.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 19 years of age at time of consent
* Have a diagnosis of RA per ACR criteria
* Must understand and voluntarily sign an informed consent form including writing consent for data protection
* Stable doses of methotrexate over the preceding 6 weeks

Exclusion Criteria:

* Pregnant or lactating females
* Previous anaphylactic response to vaccine components or to egg.
* Acute infection with T >38°C at the time of vaccination
* History of Guillain-Barre syndrome or demyelinating syndromes
* Blood transfusion within 6 months
* Any other rheumatic disease such as systemic lupus erythematosus, mixed connective tissue disease, dermatomyositis/polymyositis, and vasculitis except for secondary Sjogren's disease
* Any condition including laboratory abnormality which places the subject at unacceptable risk
* Subjects who decline to participate

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of satisfactory vaccine response | 4 weeks
  as ≥ 4-fold increase in post-vaccination titer in ≥ 2 of 4 influenza strains at 4 weeks after vaccination

SECONDARY OUTCOMES:
Proportio0n of patients who have ≥ 4-fold increase in post-vaccination titer in ≥ 3 of 4 influenza strains | 4 weeks and 16 weeks
  Proportion of patients who have ≥ 4-fold increase in post-vaccination titer in ≥ 3 of 4 influenza strains at 4 weeks and 16 weeks after vaccination
Proportion of seroprotection for each strain | 4 weeks and 16 weeks
Change from baseline in titer (in GMT) | 4 weeks and 16 weeks
Change from baseline in DAS28-4 (CRP) | 4 weeks and 16 weeks
Disease flare | 4 weeks and 16 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Park JK, Kim MJ, Choi Y, Winthrop K, Song YW, Lee EB. Effect of short-term methotrexate discontinuation on rheumatoid arthritis disease activity: post-hoc analysis of two randomized trials. Clin Rheumatol. 2020 Feb;39(2):375-379. doi: 10.1007/s10067-019-04857-y. Epub 2019 Dec 10. PMID 31823141
- [Result] Park JK, Lee YJ, Shin K, Ha YJ, Lee EY, Song YW, Choi Y, Winthrop KL, Lee EB. Impact of temporary methotrexate discontinuation for 2 weeks on immunogenicity of seasonal influenza vaccination in patients with rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2018 Jun;77(6):898-904. doi: 10.1136/annrheumdis-2018-213222. Epub 2018 Mar 23. PMID 29572291
- [Result] Park JK, Lee MA, Lee EY, Song YW, Choi Y, Winthrop KL, Lee EB. Effect of methotrexate discontinuation on efficacy of seasonal influenza vaccination in patients with rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2017 Sep;76(9):1559-1565. doi: 10.1136/annrheumdis-2017-211128. Epub 2017 May 3. PMID 28468794
- [Derived] Park JK, Lee YJ, Shin K, Kang EH, Ha YJ, Park JW, Kim MJ, Kim MH, Choi SR, Jung Y, Lee JH, In Jung J, Kim JY, Winthrop KL, Lee EB. A Multicenter, Prospective, Randomized, Parallel-Group Trial on the Effects of Temporary Methotrexate Discontinuation for One Week Versus Two Weeks on Seasonal Influenza Vaccination in Patients With Rheumatoid Arthritis. Arthritis Rheumatol. 2023 Feb;75(2):171-177. doi: 10.1002/art.42318. Epub 2022 Dec 7. PMID 35930728